CLINICAL TRIAL: NCT04935125
Title: The Effects of Combined Endurance and Strength Training on Quality of Life in Subjects With Moderate-severe Asthma: a Randomized Controlled Study.
Brief Title: The Effects of Endurance and Strength Training in Subjects With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2525CE
Record Dates: First submitted 2021-05-05; First posted 2021-06-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Asthma
Keywords: Asthma; Resistance Training; Endurance Training; Quality of Life
MeSH Terms: conditions — Asthma | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Program (Active Comparator): twelve 30-minute daily sessions of supervised incremental exercise training over a period of 3 weeks.
  Interventions: Procedure: Standard Program + Endurance and Strength training; Procedure: Standard Program
- Strength training (Experimental): twelve 30-minute daily sessions of supervised incremental exercise training over a period of 3 weeks twelve 30-minute daily sessions of supervised peripheral limb muscle training, 2 set of 6-12 repetitions
  Interventions: Procedure: Standard Program + Endurance and Strength training

INTERVENTIONS:
Procedure: Standard Program + Endurance and Strength training — Sessions of strength training added to a standard inpatient multidisciplinary programme
Procedure: Standard Program — Standard inpatient multidisciplinary programme (including endurance training)
  Arms: Standard Program

SUMMARY:
Emerging evidence suggests that regular exercise can complement medical treatment for asthma. Furthermore there are no specific recommendation on how plan exercise training. To the best of current knowledge, there isn't enough evidence of the effect of a strength training in subjects with asthma. Therefore the aim of this study is to evaluate the short and long term effects of a strength and endurance training compared with endurance training alone in subjects with asthma.

DETAILED DESCRIPTION:
To the best of current knowledge, there isn't enough evidence of the effect of a strength training in subjects with asthma. Aim of the study is evaluate the short (after pulmonary rehabilitation) and long term (after 12 months) effects of a strength and endurance training compared with endurance training alone in improving quality of life and disease control in subjects with asthma of Global Initiative for Asthma (GINA) stage from 4 to 5.This is a prospective randomized control trial. Subjects with diagnosis of asthma according to the GINA guidelines admitted to a reference centre for inpatient pulmonary rehabilitation will be randomly assigned to study or control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma step 4 to 5 under optimal medical treatment for at least 6 months according to GINA guideline
* Symptomatic despite being on treatment: Asthma Control Test (ACT) score ≥ 20 ≤24
* Able to perform and complete with studies procedures (FeNO, CPET, Six Minute Walking Test (6MWT), MVS.

Exclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) according to the Global initiative for Obstructive Lung Disease (GOLD) guidelines criteria
* Smokers or ex-smokers with pack/years ≥10
* Body Mass Index (BMI) ≥30
* Change in asthma medications in the last 30 days
* Cognitive impairment (Mini-Mental State Examination score <22)
* History of oncological, neurological, cardiovascular diseases, musculoskeletal impairment and/or medical diseases precluding exercise testing and pulmonary rehabilitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
asthma related Quality of Life | 4 weeks from enrollment
  Asthma Quality of Life Questionnaire (AQLQ). Range 0 (worst) - 7 (best)
asthma related Quality of Life | 1 year
  Asthma Quality of Life Questionnaire (AQLQ). Range 0 (worst) - 7 (best)

SECONDARY OUTCOMES:
Asthma control | 4 weeks from enrollment
  Asthma Control Questionnaire (ACQ-6). Range 0 (best) - 6 (worst)
Eosinophilic airway inflammation | 4 weeks from enrollment
  Fractional Exhaled Nitric Oxide (FeNO),
Aerobic capacity | 4 weeks from enrollment
  Maximum oxygen capacity (VO2max) assessed by Cardio Pulmonary Exercise Test, (CPET).
Quadriceps and biceps strength | 4 weeks from enrollment
  Maximal Voluntary isometric Strength (MVS).
Quadriceps and biceps strength | 1 year
  Maximal Voluntary isometric Strength (MVS).
Treatment satisfaction | 1 year
  Global Perceived Effect (GPE) score 1 (best) - 7 (worst)
Numbers of exacerbations | 1 year
  number of exacerbations in the last 12 months.
Asthma control | 1 year
  Asthma Control Questionnaire (ACQ-6) Range 0 (best) - 6 (worst)
Eosinophilic airway inflammation | 1 year
  Fractional Exhaled Nitric Oxide (FeNO).
Aerobic capacity | 1 year
  Maximum oxygen capacity(VO2max) assessed by Cardio Pulmonary Exercise Test (CPET)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Maugeri Pneumologia, Tradate, Lombardy, Italy

REFERENCES:
- [Derived] Bello GL, Oliva FM, Malovini A, Ambrosino N, Tarasconi M, Zanini A, Zampogna E. Effect of combined strength and endurance training in adults with asthma: a randomized controlled trial. J Bras Pneumol. 2025 Dec 5;51(5):e20250009. doi: 10.36416/1806-3756/e20250009. eCollection 2025. PMID 41370562